CLINICAL TRIAL: NCT05977010
Title: Evaluation of GeneXpert HIV-1 as The Gold Standard Test for HIV-1 Viral Load Count
Acronym: ProXpert
Status: Completed | Type: Observational
Sponsor: Ina-Respond (Other)
Responsible Party: Sponsor
Other Study IDs: INA104.01
Record Dates: First submitted 2018-01-11; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: HIV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a cohort study on HIV-1 patients treated in outpatient and inpatient wards of Tangerang District Hospital. The participant will be interviewed and retrieved for their demographics, treatment history, CD4 and viral load history. Blood will be drawn for HIV-1 viral load examination using Xpert® HIV-1 Viral Load [Cepheid], in-house qRT-PCR, and REALTIME HIV-1 VIRAL LOAD [Abbott]

DETAILED DESCRIPTION:
Participant candidate will be screened at Tangerang District Hospital's outpatient and inpatient units. The purpose is to get various VL values from participants with various clinical conditions (light-heavy). If a participant is willing to participate and has signed the Informed Consent Form (ICF), he/she will be interviewed for demographic data and case history (age, gender, first HIV diagnosis). After that, the participant will be physically examined (height, weight, and vital signs). Other information, such as current HIV clinical stage, current ART regimen, Viral Load value (final and highest), and CD4 (final and lowest) are collected from participant's medical records.

The participant's blood will be drawn as much as 9 ml and will be processed to obtain plasma. Plasma will be aliquoted into 3 vials for VL test using 3 devices: 1 ml using Xpert HIV-1, 1 ml using PCR (Abbott) at Dharmais Hospital, and 1 ml or leftover plasma using PCR (ABI7500) at INA-RESPOND's reference laboratory. The process follows the manufacturer's manual or the standard of sample preparation procedure and the operation of the devices at each hospital.

The result of viral load measurement will be informed to the participant via the attending physician during the participant's routine HIV treatment visit to the hospital.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive patient by the HIV Diagnoses Guideline in the Tangerang District Hospital.
* Patient older than 18 years and above.
* Willing and signed the informed consent (ICF).
* Willing to comply with the study procedures.

Exclusion Criteria:

* Suffered from a disease or having condition that could complicated the blood drawing process or increasing the risk of disease complications.
* Currently imprisoned.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of this study is 58 HIV positive patients who are currently treated in Tangerang District Hospital. Sample size is calculated based on Bland-Altman methods and 95% Confidence Interval (CI) which will be used to evaluate agreement/concordance from mean difference between three methods.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
To evaluate the performance of three different methods in measuring HIV-1 VL. | From date of patient enrolment until the date of completed result analysis for three assays, which is estimated for four (4) months.
  HIV-1 RNA concentration (copies/ml) is determined from three different plasma viral load (pVL) measurement: Xpert® HIV-1 Viral Load [Cepheid], in-house qRT-PCR observing a conserved region in HIV-1 gag gene (HXB2 1849-1896) [primer/probes: Palmer S, Wiegand AP, Maldarelli F, et al. New real-time reverse transcriptase-initiated PCR assay with single-copy sensitivity for human immunodeficiency virus type 1 RNA in plasma. J Clin Microbiol. 2003 Oct;41(10):4531-6. doi: 10.1128/JCM.41.10.4531-4536.2003. PMID: 14532178; PMCID: PMC254331], and REALTIME HIV-1 VIRAL LOAD [Abbott].

SECONDARY OUTCOMES:
To evaluate correlation of HIV-1 pVL measurement using Xpert® HIV-1 Viral Load [Cepheid] and in-house qRT-PCR [HIV-1 gag gene (HXB2 1849-1896), Palmer S, Wiegand AP, Maldarelli F, et al. J Clin Microbiol. 2003 Oct;41(10):4531-6] | From date of patient enrolment until the date of completed result analysis for three assays, which is estimated for four (4) months.
  Mean difference of HIV-1 RNA concentration.
To evaluate correlation of HIV-1 pVL measurement using Xpert® HIV-1 Viral Load [Cepheid] and REALTIME HIV-1 VIRAL LOAD [Abbott]. | From date of patient enrolment until the date of completed result analysis for three assays, which is estimated for four (4) months.
  Mean difference of HIV-1 RNA concentration.
To evaluate correlation and mean difference in HIV-1 pVL measurement using REALTIME HIV-1 VIRAL LOAD [Abbott] and in-house qRT-PCR [HIV-1 gag gene (HXB2 1849-1896), Palmer S, Wiegand AP, Maldarelli F, et al. J Clin Microbiol. 2003 Oct;41(10):4531-6]. | From date of patient enrolment until the date of completed result analysis for three assays, which is estimated for four (4) months.
  Mean difference of HIV-1 RNA concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. dr. Tuti Parwati Merati, Sp.PD.KPTI, Principal Investigator — Ina-Respond
Locations (1):
- RSU Kabupaten Tangerang, Tangerang, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No